CLINICAL TRIAL: NCT01818635
Title: Phase 4 Study of to Investigation the Effect of Montelukast on Behavior Problems in Children With Asthma
Brief Title: To Investigate the Effect of Montelukast on Behavior Problems in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Fatih University (Other)
Collaborators: Kecioren Teaching and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Ahmet Z. Akelma, Fatih University Medical School, Fatih University
Other Study IDs: FK-0663
Record Dates: First submitted 2013-03-22; First posted 2013-03-26 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Asthma, Behavior Problem, Montelukast
MeSH Terms: conditions — Asthma; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study to investigate whether montelukast lead to behavior problems in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* To have asthmatic children aged 18-60 months
* To have that receive prophylactic treatment for asthma
* Healthy children will be enrolled among those being brought for routine controls

Exclusion Criteria:

* Children with other chronic disease
* Children with chronic drug use (except for the treatment of asthma)

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We planned to include who who treated for asthmatic children and healthy controls in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of montelukast on behavior problems in children with asthma | 8 months
  Montelukast frequently used in the treatment of asthmatic children. However, we believe that montelukast lead to behavior problems. In this study, we aimed to investigate that intake of montelukast whether lead to behavior problems.

SECONDARY OUTCOMES:
To compare the effects of inhaled corticosteroids and montelukast on the behavior problems. | 8 months
  In this study, it will be compared the effect on behavior changes between intake of inhaled steroid and montelukast.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Fatih University Medical School, Ankara
  - Fatih University, Ankara